CLINICAL TRIAL: NCT05671614
Title: Skeletal Muscle Regeneration in Survivors of Critical Illness: How to Prevent Satellite Cell Failure?
Acronym: SATELLITE
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Adéla Krajčová, MD, PhD, Principal Investigator, Charles University, Czech Republic
Other Study IDs: NU21J-06-00078
Record Dates: First submitted 2022-08-16; First posted 2023-01-04 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Intensive Care Unit-acquired Weakness
Keywords: intensive care unit-acquired weakness; critically ill; skeletal muscle regeneration; satellite cells
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critically ill patients: Critically ill patients with sudden onset of disease receiving mechanical ventilation, to be enrolled within 72 hours of admission, who are likely to need 7 days or more of ICU stay.
- Volunteers with a very good to excellent performance status: Elective hip surgery patients with a very good to excellent performance status, only limited to joint pain (ECOG 0)

SUMMARY:
Modern intensive care enables patients to survive insults that in the past would have been supralethal. Nonetheless, increased number of survivors suffer from failed functional outcomes associated with prolonged muscle weakness and fatiguability. Whilst alterations of skeletal muscle biology that occur during critical illness slowly disappear over the period of months, muscle weakness remains. Recent pilot studies have shown that muscle weakness is associated with loss and alteration of satellite skeletal muscle cells, which are supposed to proliferate and repair damaged muscle tissue. The pathogenesis of this phenomenon has not been fully understood. In this grant project, we will study function and structure of satellite cells and their organelles (particularly mitochondria) using both classical bioenergetics and advanced microscopic techniques. Satellite cells will be isolated from biopsies taken from critically ill patients with developed muscle weakness in the acute and protracted phase of a disease and after 6 months. In time points, an ultrasound examination of muscle mass will be performed, and metabolism will be assessed using insulin clamps. In an in vitro experiments, we will test also effect of nutritional and anabolic factors and drugs, commonly used in ICU, on satellite cells. In a control branch, cells will be isolated from skeletal muscle of volunteers undergoing elective hip replacement surgery. Results of this study could significantly contribute to understanding of mechanisms leading to ICU acquired muscle weakness and to identify therapeutic strategy in future.

DETAILED DESCRIPTION:
Background:

Muscle weakness is a common complication in patients who survived a serious critical illness or trauma. Altered muscle strength and functional ability significantly worsens the patients' performance and quality of life. Specific treatment does not exist and the pathogenesis is not yet fully understood. Acute sepsis or extensive inflammatory response are the main risk factors for the muscle weakness development in critically ill patients. Recent studies have shown that muscle weakness can be caused by the loss of ability of skeletal muscle cells to react to the injury and regenerate. Skeletal muscle satellite cells, which are localized beneath the basal lamina of individual muscle fibers, are responsible for muscle regeneration. After the muscle damage, satellite cells are activated from quiescent state (G0 phase) and enter the cell cycle (G1 phase). Subsequently, they proliferate and differentiate into the myoblasts which then fuse and form multinucleated cylindrical myotubes. The cells then merge into the myofibrils and join the muscle fibers that were not damaged. Some satellite cells return to the G0 state to replenish the pool of quiescent skeletal muscle cells. In response to satellite cell damage, mitochondrial biogenesis and synthesis of new myofibrillar proteins are activated to build the new muscle mass containing new intracellular content. Thus, satellite cells have a crucial role for muscle fiber regeneration. Pilot studies performed on animal models (e. g. laboratory mice that developed the acute sepsis) demonstrated a reduction in mitochondrial content and DNA, increased production of reactive oxygen species and changes in oxidative phosphorylation. The abnormalities in the bioenergetic profile of satellite cells are considered a cause of their reduced ability to regenerate. However, the exact mechanism has not yet been fully elucidated. Changes in the mitochondrial structure and dynamics of satellite cells in critically ill patients are also unknown. In last years, the association of mitochondrial functions with mitochondrial dynamics has been investigated in various pathological conditions and diseases. Depending on external insults and metabolic demands, mitochondria undergo dramatic shape changes that can have a very significant impact on cellular metabolism. The balanced process of mitochondrial fission and fusion plays a key role in the mitochondrial biogenesis and removal of damaged mitochondria. The process is absolutely necessary for the proper growth and function of the muscle tissue. Mitochondrial dynamics and morphology can be altered under pathological circumstances: under the mild stress and starvation, mitochondrial morphology can change from small spheres or short rods to long tubules with an increased capacity for oxidative phosphorylation. On the other hand, acute severe stress leads to a mitochondrial fission and defective oxidative phosphorylation. Several studies performed on animal models demonstrated that proteins responsible for the process of mitochondrial fusion and fission are absolutely crucial for the proper growth and function of skeletal muscle cells. Therefore, alterations in mitochondrial dynamics often play a crucial role in skeletal muscle dysfunction and have been recently extensively studied in several myopathies.

In this project, the investigators would like to investigate the causal relationships between mitochondrial function and their shape in satellite cells obtained from critically ill patients in the acute, protracted and post-ICU phase of critical illness.

Hypotheses and aims of the project:

In light of this, the investigators hypothesize that critical illness induces damage to satellite cells in skeletal muscle that later impairs skeletal muscle structural and functional recovery and contributes to persistent weakness and failed functional outcome.

First, structural and functional (incl. bioenergetic) characteristics of satellite cells will be compared in acute, protracted and post-ICU phase in critically ill patients vs. control subjects. Second, the investigators will test the hypothesis that structural and/or functional alteration of satellite cells corelate with gross muscle mass and power in survivors of critical illness. Third, the factors that influence bioenergetics and mitochondrial morphology of satellite cells will be studied (such as extracellular inflammatory milieu, drugs common in ICU as well as nutritional and anabolic factors).

Design:

Prospective cohort study with exploratory physiological end-points.

Study subjects:

Critically ill patients: receiving mechanical ventilation to be enrolled within 72 hours of admission, who are likely to need 7 days or more of ICU stay; sudden onset of disease, which can be determined in time (such as trauma, stroke, sudden cardiac arrest etc.).

Control subjects: orthopedic patients undergoing elective hip replacement surgery with a very good to excellent performance status, only limited to joint pain (ECOG 0).

Informed consent procedure:

All patients with capacity will be asked to provide a prospective written informed consent. For patients without capacity, a deferred consent procedure will take a place. In this case, an independent clinician will review and sign that the patient is lacking capacity and he/she fulfills all criteria to be enrolled to the study. The patient's next of kin will be informed about the study as soon as practical with the aid of information leaflet. The patient will be asked to provide and sign informed consent as soon as he/she regains the capacity to do so. In case of consent refusal, patient's data will not be used in per-protocol analysis.

Methods:

General methodological approaches to be used are as follows. Time points: Eligible patients will be assessed at the baseline, after 7 days and after 6 months by clinical tests, metabolic tests and muscle biopsies. Briefly, on day 0 muscle mass will be assessed using diagnostic ultrasound (a measurement of rectus muscle cross-sectional area) and biopsy of musculus vastus lateralis will be performed using Bergström needle. Baseline blood samples will be taken, plasma will be separated and frozen at -80° C for the later analysis of cytokines and hormone levels. Urine samples will be collected daily, surfaced with toluene and stored in a deep freeze facility for later determination of nitrogen content and 3-methyl histidine levels (to calculate muscle catabolism rate and nitrogen balance). On day 7, all above mentioned procedures will be performed again. In addition, whenever the patient regains consciousness, also muscle power by Medical Research Council (MRC) score will be assessed (standardized testing of muscle power [0-5] on 12 muscle groups on all 4 limbs, giving the score 0-60 (60 suggesting normal muscle power)). At ICU discharge, the patients and relatives will be asked to provide contact details for 6 months follow up. On day 180, all the procedures will be repeated. Furthermore, insulin sensitivity will be measured after overnight fasting by hyperinsulinaemic euglycemic clamp on days 7 and 180.

Clinical outcomes: will be assessed by objective validated tests such as SF-36 questionnaire for the quality of life assessment, Medical Research Council Score of muscle power and 6-minutes walking test to measure aerobic performance.

Metabolic characteristics: will be assessed at the whole body level by hyperinsulinaemic euglycaemic clamps and at the tissue level by vastus lateralis biopsies. Insulin sensitivity and substrate oxidation will be measured after overnight fasting by hyperinsulinaemic euglycemic clamp.

Laboratory procedures: mitochondrial research: muscle tissue biopsies will be performed from vastus lateralis muscle by Bergström needle biopsy technique. The sample from each biopsy will be separated into three parts (from 25-100mg per each). One part will be immediately frozen in liquid nitrogen-cooled isopentane for later analysis of muscle fibres typing and immunohistochemistry analysis. The second part will be placed into the respiration medium on ice for the preparation of homogenates and measurement on high-resolution respirometry which enables to determine the function of individual respiratory complexes in the cytosolic context and measure basic functional metabolic indices. Mainly, ATP production, mitochondrial uncoupling, electron transport chain capacity and respiration linked to individual complexes will be assessed. The third part will be used for isolation and culture of skeletal muscle cells. Firstly, satellite cells from biopsies using FACS or magnetic beads will be isolated. The satellite cells will be cultivated and global mitochondrial indices will be assessed by measurement of oxygen consumption rate. This will be processed with extracellular flux analyzer or high resolution respirometry which enables measurement of oxygen consumption rate and lactate production in a real time. This enables to determine ATP production in living cells, uncoupling of inner mitochondrial membrane, maximal respiratory capacity of respiratory chain, glycolytic capacity and fatty acid oxidation or respiration linked to individual complexes of respiratory chain. Simultaneously, reactive oxygen species and mitochondrial membrane potential will be measured. Additionally, shape and size of mitochondria, density of mitochondrial network and dynamic arrangement of these interconnected organelles will be analyzed using confocal laser scanning microscopy in live-cell imaging. All the parameters will be studied in the acute, protracted and post-ICU phase of critical illness.

ELIGIBILITY:
Eligibility Criteria for group of Critically ill patients:

Inclusion Criteria:

* Critically ill patients receiving mechanical ventilation, to be enrolled within 72 hours of admission, who are likely to need 7 days or more of ICU stay
* Sudden onset of disease, which can be determined in time (such as trauma, stroke, sudden cardiac arrest etc.)
* Informed consent signed by patient or patient's representative

Exclusion Criteria:

* Unlikely to survive 6 months
* Premorbid downslope functional trajectory or poor performance status (ECOG Gr. 3 or worse) or baseline functional status unknown
* Bleeding disorder (INR≥1.5 or PLT< that would preclude muscle biopsies)
* Known mitochondrial disease
* Endocrine crisis as a reason for admission
* Pregnant women

Eligibility Criteria for a control group:

Elective hip surgery patients with a very good to excellent performance status, only limited to joint pain (ECOG 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sudden onset of disease receiving mechanical ventilation, to be enrolled within 72 hours of admission, who are likely to need 7 days or more of ICU stay. Study population will be compared with control group consisting of patients undergoing hip replacement surgery with a very good to excellent performance status.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life as per 36-Item Short Form Health Survey (SF-36) | on day 180
  A set of quality-of-life measures. A questionnaire includes questions about: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The minimum and maximum scores are 0 and 100. A higher score defines a more favorable health state.
Changes of muscle mass between baseline, day 7 and day 180 | Changes between days 0, 7 and 180
  By measurement of musculus rectus femoris cross-sectional area by diagnostic ultrasound.
A measurement of muscle power by Medical Research Council Score | on day 180 (eventually on day 7 if the patient is conscious)
  A standardized testing of muscle power [0-5] on 12 muscle groups on all 4 limbs using Medical Research Council Score, giving the score from minimum 0 to maximum 60. A higher score defines a more favorable health state, 60 points suggest a normal muscle power.
Changes of mitochondrial function of satellite cells between baseline, day 7 and day 180 | Changes between days 0, 7 and 180
  Mitochondrial functional parameters will be assessed by Extracellular XF24 Seahorse Analyzer or high-resolution respirometry which enables continous real-time measurement of oxygen consumption in living cells at the baseline and after addition of various substrates, uncouplers and inhibitors of the respiratory chain. This allow to estimate parameters as ATP production, maximal respiratory capacity, respiration in baseline etc. The techniques measure oxygen consumption rate of living cells in pmol/min.
Changes of mitochondrial structure of satellite cells between baseline, day 7 and day 180 | Changes between days 0, 7 and 180
  A mitochondrial structure and architecture of its network (mitochondrial density and a length of its branches etc.) will be assessed after staining of mitochondria by fluorescent probes and imaging on confocal laser scanning microscopy. The length/density will be measured in microns/microns 2.

SECONDARY OUTCOMES:
Nitrogen balance measured in g/m2 of body surface area | on first 7 days
  From collected urine samples, a determination of nitrogen content and 3-methyl histidine levels will be performed (to calculate muscle catabolism rate and nitrogen balance).
6-minutes walking test to measure aerobic performance | on day 180
  6-minutes of exercise (walking) test used to assess aerobic capacity and endurance.
Changes of insulin sensitivity between days 7 and 180 | Changes between days 7 and 180
  This parameter will be measured after overnight fasting by hyperinsulinaemic euglycemic clamp.
Length of ICU stay in days | on day 28
  A number of days spent on ICU.
Number of ventilator-free days | on day 28
  A number of ventilator-free days spent on ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from de-identified individual patients will be made available in a public database.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Hermans G, Van den Berghe G. Clinical review: intensive care unit acquired weakness. Crit Care. 2015 Aug 5;19(1):274. doi: 10.1186/s13054-015-0993-7. PMID 26242743
- [Background] Horn J, Hermans G. Intensive care unit-acquired weakness. Handb Clin Neurol. 2017;141:531-543. doi: 10.1016/B978-0-444-63599-0.00029-6. PMID 28190434
- [Background] Powers SK, Lynch GS, Murphy KT, Reid MB, Zijdewind I. Disease-Induced Skeletal Muscle Atrophy and Fatigue. Med Sci Sports Exerc. 2016 Nov;48(11):2307-2319. doi: 10.1249/MSS.0000000000000975. PMID 27128663
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] Dos Santos C, Hussain SN, Mathur S, Picard M, Herridge M, Correa J, Bain A, Guo Y, Advani A, Advani SL, Tomlinson G, Katzberg H, Streutker CJ, Cameron JI, Schols A, Gosker HR, Batt J; MEND ICU Group; RECOVER Program Investigators; Canadian Critical Care Translational Biology Group. Mechanisms of Chronic Muscle Wasting and Dysfunction after an Intensive Care Unit Stay. A Pilot Study. Am J Respir Crit Care Med. 2016 Oct 1;194(7):821-830. doi: 10.1164/rccm.201512-2344OC. PMID 27058306
- [Background] Zammit PS, Relaix F, Nagata Y, Ruiz AP, Collins CA, Partridge TA, Beauchamp JR. Pax7 and myogenic progression in skeletal muscle satellite cells. J Cell Sci. 2006 May 1;119(Pt 9):1824-32. doi: 10.1242/jcs.02908. Epub 2006 Apr 11. PMID 16608873
- [Background] Schultz E, McCormick KM. Skeletal muscle satellite cells. Rev Physiol Biochem Pharmacol. 1994;123:213-57. doi: 10.1007/BFb0030904. PMID 8209136
- [Background] Monge C, DiStasio N, Rossi T, Sebastien M, Sakai H, Kalman B, Boudou T, Tajbakhsh S, Marty I, Bigot A, Mouly V, Picart C. Quiescence of human muscle stem cells is favored by culture on natural biopolymeric films. Stem Cell Res Ther. 2017 May 2;8(1):104. doi: 10.1186/s13287-017-0556-8. PMID 28464938
- [Background] Bentzinger CF, Wang YX, Rudnicki MA. Building muscle: molecular regulation of myogenesis. Cold Spring Harb Perspect Biol. 2012 Feb 1;4(2):a008342. doi: 10.1101/cshperspect.a008342. PMID 22300977
- [Background] Yin H, Price F, Rudnicki MA. Satellite cells and the muscle stem cell niche. Physiol Rev. 2013 Jan;93(1):23-67. doi: 10.1152/physrev.00043.2011. PMID 23303905
- [Background] Sin J, Andres AM, Taylor DJ, Weston T, Hiraumi Y, Stotland A, Kim BJ, Huang C, Doran KS, Gottlieb RA. Mitophagy is required for mitochondrial biogenesis and myogenic differentiation of C2C12 myoblasts. Autophagy. 2016;12(2):369-80. doi: 10.1080/15548627.2015.1115172. PMID 26566717
- [Background] Pham AH, McCaffery JM, Chan DC. Mouse lines with photo-activatable mitochondria to study mitochondrial dynamics. Genesis. 2012 Nov;50(11):833-43. doi: 10.1002/dvg.22050. Epub 2012 Aug 11. PMID 22821887
- [Background] Wagatsuma A, Sakuma K. Mitochondria as a potential regulator of myogenesis. ScientificWorldJournal. 2013;2013:593267. doi: 10.1155/2013/593267. Epub 2013 Feb 3. PMID 23431256
- [Background] Chen H, Vermulst M, Wang YE, Chomyn A, Prolla TA, McCaffery JM, Chan DC. Mitochondrial fusion is required for mtDNA stability in skeletal muscle and tolerance of mtDNA mutations. Cell. 2010 Apr 16;141(2):280-9. doi: 10.1016/j.cell.2010.02.026. PMID 20403324
- [Background] Mohiuddin M, Lee NH, Moon JY, Han WM, Anderson SE, Choi JJ, Shin E, Nakhai SA, Tran T, Aliya B, Kim DY, Gerold A, Hansen LM, Taylor WR, Jang YC. Critical Limb Ischemia Induces Remodeling of Skeletal Muscle Motor Unit, Myonuclear-, and Mitochondrial-Domains. Sci Rep. 2019 Jul 2;9(1):9551. doi: 10.1038/s41598-019-45923-4. PMID 31266969
- [Background] Krajcova A, Ziak J, Jiroutkova K, Patkova J, Elkalaf M, Dzupa V, Trnka J, Duska F. Normalizing glutamine concentration causes mitochondrial uncoupling in an in vitro model of human skeletal muscle. JPEN J Parenter Enteral Nutr. 2015 Feb;39(2):180-9. doi: 10.1177/0148607113513801. Epub 2013 Nov 29. PMID 24291738
- [Background] Jiroutkova K, Krajcova A, Ziak J, Fric M, Gojda J, Dzupa V, Kalous M, Tumova J, Trnka J, Duska F. Mitochondrial Function in an In Vitro Model of Skeletal Muscle of Patients With Protracted Critical Illness and Intensive Care Unit-Acquired Weakness. JPEN J Parenter Enteral Nutr. 2017 Sep;41(7):1213-1221. doi: 10.1177/0148607116657649. Epub 2016 Jun 29. PMID 27358332
- [Background] Krajcova A, Lovsletten NG, Waldauf P, Fric V, Elkalaf M, Urban T, Andel M, Trnka J, Thoresen GH, Duska F. Effects of Propofol on Cellular Bioenergetics in Human Skeletal Muscle Cells. Crit Care Med. 2018 Mar;46(3):e206-e212. doi: 10.1097/CCM.0000000000002875. PMID 29240609
- [Background] Urban T, Waldauf P, Krajcova A, Jiroutkova K, Halacova M, Dzupa V, Janousek L, Pokorna E, Duska F. Kinetic characteristics of propofol-induced inhibition of electron-transfer chain and fatty acid oxidation in human and rodent skeletal and cardiac muscles. PLoS One. 2019 Oct 4;14(10):e0217254. doi: 10.1371/journal.pone.0217254. eCollection 2019. PMID 31584947
- [Background] Aguer C, Foretz M, Lantier L, Hebrard S, Viollet B, Mercier J, Kitzmann M. Increased FAT/CD36 cycling and lipid accumulation in myotubes derived from obese type 2 diabetic patients. PLoS One. 2011;6(12):e28981. doi: 10.1371/journal.pone.0028981. Epub 2011 Dec 16. PMID 22194967
- [Background] Kuznetsov AV, Kehrer I, Kozlov AV, Haller M, Redl H, Hermann M, Grimm M, Troppmair J. Mitochondrial ROS production under cellular stress: comparison of different detection methods. Anal Bioanal Chem. 2011 Jun;400(8):2383-90. doi: 10.1007/s00216-011-4764-2. Epub 2011 Feb 20. PMID 21336935
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Ziak J, Krajcova A, Jiroutkova K, Nemcova V, Dzupa V, Duska F. Assessing the function of mitochondria in cytosolic context in human skeletal muscle: adopting high-resolution respirometry to homogenate of needle biopsy tissue samples. Mitochondrion. 2015 Mar;21:106-12. doi: 10.1016/j.mito.2015.02.002. Epub 2015 Feb 17. PMID 25701243
- [Background] Jiroutkova K, Krajcova A, Ziak J, Fric M, Waldauf P, Dzupa V, Gojda J, Nemcova-Furstova V, Kovar J, Elkalaf M, Trnka J, Duska F. Mitochondrial function in skeletal muscle of patients with protracted critical illness and ICU-acquired weakness. Crit Care. 2015 Dec 24;19:448. doi: 10.1186/s13054-015-1160-x. PMID 26699134
- [Derived] Genserova L, Duska F, Krajcova A. beta-hydroxybutyrate exposure restores mitochondrial function in skeletal muscle satellite cells of critically ill patients. Clin Nutr. 2024 Jun;43(6):1250-1260. doi: 10.1016/j.clnu.2024.04.009. Epub 2024 Apr 9. PMID 38653008

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT05671614/Prot_ICF_000.pdf